CLINICAL TRIAL: NCT07390903
Title: Global Longitudinal Strain as a Predictor of Difficult Separating From Cardiopulmonary Bypass
Brief Title: GLS in Difficult CPB Weaning
Status: Recruiting | Type: Observational
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Collaborators: University of Rome Tor Vergata (Other); San Raffaele University Hospital, Italy (Other)
Responsible Party: Principal Investigator, mustafa emre gürcü, Attending Medical Doctor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2025/14/1189
Record Dates: First submitted 2026-01-12; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiopulmonary Bypass; Coronary Artery Bypass; Heart Valve Diseases; Echocardiography; Intraoperative Complications; Postoperative Complications (Cardiopulmonary)
MeSH Terms: conditions — Heart Valve Diseases; Intraoperative Complications; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Easy CPB Separation: Easy separation from CPB was defined as no pharmacologic support or use of a single agent (either vasoactive or inotropic).
  Interventions: Diagnostic Test: Myocardial strain imaging
- Difficult CPB Separation: Difficult CPB separation can be defined as the need of at least 2 inotropes or vasopressors to successfully accomplish the separation from CPB.
  Interventions: Diagnostic Test: Myocardial strain imaging

INTERVENTIONS:
Diagnostic Test: Myocardial strain imaging — Two-dimensional strain analysis was performed using frame-by-frame tracking of unique patterns of bright and dark pixels in grayscale (B-mode) sector images to assess myocardial deformation. The frame rate was maintained between 40 and 90 Hz. The myocardium in each image was divided into six myocardial segments, which were individually assessed for tracking quality. GLS was calculated as the average strain value of 18 myocardial segments obtained from the three echocardiographic views. Patients were included in the final analysis if at least 15 out of 18 segments were considered acceptable for strain measurement by the investigator.

SUMMARY:
The goal of this observational study is to learn whether global longitudinal strain (GLS), measured by echocardiography, can predict difficulty separating from cardiopulmonary bypass (CPB) in adults undergoing elective cardiac surgery.

The main questions it aims to answer are:

* Can preoperative GLS measurement predict difficult separation from CPB?
* Are GLS values associated with outcomes such as intensive care unit (ICU) stay, hospital stay, cardiac biomarkers, or 30-day mortality?

Participants will:

* Undergo standard cardiac surgery requiring CPB
* Have echocardiographic assessments (TTE before and after surgery)
* Have their recovery and outcomes monitored, including ICU and hospital stay, postoperative labs, and survival within 30 days

DETAILED DESCRIPTION:
Background and Rationale

Difficult separation from cardiopulmonary bypass (CPB) is a serious intraoperative complication associated with increased perioperative morbidity and mortality. Myocardial contractility is the key determinant of successful CPB separation, and perioperative echocardiography is an established method for evaluating ventricular function. Conventionally, left ventricular ejection fraction (LVEF) measured by Simpson's biplane method is used to assess myocardial performance. However, LVEF has notable limitations, including high inter-operator variability, preload/afterload dependence, and poor sensitivity in detecting early myocardial dysfunction.

Global longitudinal strain (GLS), measured by two-dimensional speckle-tracking echocardiography, has emerged as a sensitive, reproducible, and geometry-independent parameter of myocardial function. GLS can detect subtle ventricular dysfunction earlier than conventional LVEF and has demonstrated prognostic value in a variety of clinical settings. Despite this, its use in the perioperative cardiac surgery population remains limited, partly due to uncertainty about the optimal timing of assessment. Anesthesia induction, CPB, and myocardial protection strategies may alter myocardial performance, and therefore both absolute GLS values and dynamic perioperative changes may carry prognostic significance.

Study Objectives

The primary objective of this prospective, multicenter, observational study is to evaluate the predictive value of GLS measurements for difficult separation from CPB. Specifically, the study will assess whether GLS measured by preoperative transthoracic echocardiography (TTE) can independently predict the need for multiple inotropic/vasoactive agents during CPB weaning.

Secondary objectives include exploring the associations between GLS parameters and postoperative outcomes such as intensive care unit (ICU) and hospital length of stay, postoperative changes in cardiac biomarkers, and all-cause 30-day mortality.

Methods

Eligible patients are adults (>18 years) scheduled for elective cardiac surgery requiring CPB, including isolated valve replacement or repair, coronary artery bypass grafting (CABG), combined procedures, and ascending aortic/arch surgery. Patients undergoing emergency or redo surgery, those with contraindications to TEE, or in critical preoperative states (mechanical circulatory support, inotrope dependence, atrial fibrillation, or mechanical ventilation) are excluded.

Echocardiographic assessments are performed at standardized time points: preoperative TTE (T1), intraoperative TEE after induction (T2, if performed), before CPB initiation (T3), immediately after CPB weaning (T4), and following sternal closure (T5). Intraoperative TEE is not mandated by the protocol but may be performed according to institutional practice or operator discretion. GLS analysis follows American Society of Echocardiography (ASE) guidelines, averaging strain from 18 myocardial segments.

Anesthetic and surgical protocols follow institutional standards, with cardioplegia delivered via Buckberg's or del Nido solutions. Clinical, intraoperative, and postoperative data-including operative times, need for pharmacologic support, and recovery variables-are collected systematically by trained staff.

Outcomes

* Primary Endpoint: Ability of GLS value to predict difficult CPB separation, defined as the need for at least two vasoactive or inotropic agents.
* Secondary Endpoints: Association of GLS with ICU/hospital length of stay, postoperative biomarker trends, hospital readmission, and all-cause mortality within 30 days.

Significance

This study addresses a clinically important knowledge gap by evaluating the GLS as a novel predictor of intraoperative difficulty and adverse outcomes in cardiac surgery. If validated, GLS assessment could enhance perioperative risk stratification, guide intraoperative decision-making, and ultimately improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years.
* Scheduled for elective cardiac surgery requiring cardiopulmonary bypass (CPB).
* Provided written informed consent to participate.
* Eligible surgical procedures include:

  * Isolated mitral valve replacement or repair.
  * Isolated aortic valve replacement or repair.
  * Isolated coronary artery bypass grafting (CABG).
  * Combined valve and CABG surgery.
  * Multiple valve replacement or repair.
  * Surgery involving the ascending aorta or aortic arch.

Exclusion Criteria

* Emergency cardiac surgery.
* Redo cardiac surgery.
* Contraindications to transesophageal echocardiography (TEE).
* Critical preoperative conditions, including:

  * Ongoing inotropic drug therapy.
  * Preoperative mechanical circulatory support (e.g., IABP, ECMO, VAD).
  * Requirement for mechanical ventilation.
  * Preoperative atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective cardiac surgery requiring cardiopulmonary bypass at participating tertiary cardiac surgery centers. The study recruits participants from routine surgical practice in academic and high-volume referral hospitals, where both valve and coronary artery procedures are performed. Consecutive eligible patients who provide informed consent are enrolled prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the predictive value of GLS measurements for difficult separation from cardiopulmonary bypass. | perioperative
  Separating from CPB was categorized as easy and difficult separation from CPB. Easy separation from CPB was defined as no pharmacologic support or use of a single agent (either vasoactive or inotropic). Difficult CPB separation can be defined as the need of at least 2 inotropes or vasopressors to successfully accomplish the separation from CPB

SECONDARY OUTCOMES:
To assess the associations between strain imaging and ICU/hospital length of stay, postoperative trajectories of cardiac biomarkers, and all-cause mortality. | Post operative 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- University of Rome Tor Vergata, Rome, Italy
- Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monaco F, Di Prima AL, Kim JH, Plamondon MJ, Yavorovskiy A, Likhvantsev V, Lomivorotov V, Hajjar LA, Landoni G, Riha H, Farag AMGA, Gazivoda G, Silva FS, Lei C, Bradic N, El-Tahan MR, Bukamal NAR, Sun L, Wang CY. Management of Challenging Cardiopulmonary Bypass Separation. J Cardiothorac Vasc Anesth. 2020 Jun;34(6):1622-1635. doi: 10.1053/j.jvca.2020.02.038. Epub 2020 Feb 29. PMID 32276758
- [Background] Benson MJ, Silverton N, Morrissey C, Zimmerman J. Strain Imaging: An Everyday Tool for the Perioperative Echocardiographer. J Cardiothorac Vasc Anesth. 2020 Oct;34(10):2707-2717. doi: 10.1053/j.jvca.2019.11.035. Epub 2019 Dec 7. PMID 31919005
- [Background] Sonny A, Alfirevic A, Sale S, Zimmerman NM, You J, Gillinov AM, Sessler DI, Duncan AE. Reduced Left Ventricular Global Longitudinal Strain Predicts Prolonged Hospitalization: A Cohort Analysis of Patients Having Aortic Valve Replacement Surgery. Anesth Analg. 2018 May;126(5):1484-1493. doi: 10.1213/ANE.0000000000002684. PMID 29200066
- [Background] Chan PG, Seese L, Aranda-Michel E, Sultan I, Gleason TG, Wang Y, Thoma F, Kilic A. Operative mortality in adult cardiac surgery: is the currently utilized definition justified? J Thorac Dis. 2021 Oct;13(10):5582-5591. doi: 10.21037/jtd-20-2213. PMID 34795909
- [Background] Denault AY, Tardif JC, Mazer CD, Lambert J; BART Investigators. Difficult and complex separation from cardiopulmonary bypass in high-risk cardiac surgical patients: a multicenter study. J Cardiothorac Vasc Anesth. 2012 Aug;26(4):608-16. doi: 10.1053/j.jvca.2012.03.031. Epub 2012 May 11. PMID 22578975